CLINICAL TRIAL: NCT06936774
Title: Improving Functional Outcomes and Quality of Life in Patients With Rectal Cancer After Surgery With Intensified Follow-up & Surveillance - a Randomized Controlled Trial (iRECOVER)
Brief Title: Improving Functional Outcomes and Quality of Life in Patients With Rectal Cancer After Surgery With Intensified Follow-up & Surveillance
Acronym: iRECOVER
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: St. Claraspital AG (Other); Clarunis - Universitäres Bauchzentrum Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRECOVER_2025
Record Dates: First submitted 2025-03-24; First posted 2025-04-20 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: LARS - Low Anterior Resection Syndrome; Rectal Cancer Surgery; Rectal Cancer; Quality of Life (QOL)
Keywords: LARS; Low Anterior Resection Syndrome; Intensified follow-up; Rectal cancer; Rectal resection; Low anterior resection
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Intervention group: Intensified follow-up program consisting of of several follow-up visits and medical treatment, pelvic floor muscle training and gynaecological and urological co-treatment in case of LARS symptoms and urinary or sexual complaints which will be recorded using questionnaires.
  Control group: Treatment according to standard, recording of symptoms using questionnaires only at beginning and end of the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intensified follow-up program consisting of of several follow-up visits at 1, 4, 7 and 13 months and medical treatment, pelvic floor muscle training and gynaecological and urological co-treatment in case of LARS symptoms and urinary or sexual complaints which will be recorded using questionnaires.
  Interventions: Other: Intensified follow-up program
- Control group (No Intervention): Treatment according to standard guidelines, recording of symptoms using questionnaires at 1 and 13 months.

INTERVENTIONS:
Other: Intensified follow-up program — The study intervention will be an intensified follow-up program which consists of different measures. Patients will attend follow-up visits 1, 4, 7 and 13 months after ileostomy repositioning, at which LARS symptoms, quality of life as well as sexual and urinary function will be recorded using various questionnaires. In case of LARS symptoms patients will receive medical treatment with loperamide and metamucil as well as pelvic floor muscle training (including biofeedback and home exercises). Regarding pelvic floor muscle training we are planning nine sessions instructed by physiotherapy staff. In case of therapy-resistant LARS symptoms after 6 months sacral neurostimulation is offered to the patients with a focus on incontinence symptoms and desire for surgery or transanal irrigation in patients with a focus on voiding disorders. In case of urinary and sexual complaints patients are referred to our urology or gynaecology department for further diagnostic and treatment.
  Arms: Intervention group

SUMMARY:
The goal of this clinical study is to gain further insights into the treatment of patients with Low Anterior Resection Syndrome (LARS) symptoms after rectal resection. The main question is: Can LARS symptoms and quality of life be improved by implementing an intensified follow-up program? Researchers will compare the results of the intervention group with the results of a control group in which patients do not receive an intensified follow-up program to determine whether the intervention works. Participants will undergo an intensified follow-up program which consists of several follow-up visits and medical treatment, pelvic floor muscle training and gynaecological and urological co-treatment in case of LARS symptoms and urinary or sexual complaints.

DETAILED DESCRIPTION:
Background: After surgical treatment of patients with rectal cancer, up to 65% experience a symptom complex known as LARS (Low Anterior Resection Syndrome). Those affected suffer from symptoms such as fecal incontinence, frequent bowel movements and a strong urge to defecate, which can severely impair their quality of life. Therapy options include treatment with medication such as bulking agents or drugs that reduce bowel motility, pelvic floor muscle training or stimulation of the nerves that control the function of the rectum and pelvic floor.

Objective: The aim of the present study is to investigate whether an intensified follow-up program can improve the LARS symptoms and consequently the quality of life of patients after rectal resection. If the planned study shows success of the program, we will be able to structurally improve the aftercare of those affected.

Methods: The study is being conducted at several centers in Switzerland, including St. Claraspital Basel. Patients who have had a rectal resection are recruited prior to the repositioning of the artificial bowel outlet, which was created during the primary operation, and randomly assigned to one of the both study groups (intensified follow-up or standard treatment). The symptoms are recorded using various questionnaires and patients will be treated according to our action plan. If LARS symptoms occur, patients receive drug treatment, pelvic floor physiotherapy and, if necessary, sacral neurostimulation, which means implanting a device which stimulates the nerves that control the function of the rectum and pelvic floor. If patients suffer from urinary problems or impaired sexual function they will be referred to our urology or gynecology department for further diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years
* patients with rectal cancer in the middle and lower third of the rectum in stages I to IV who underwent LAR with TME and protective ileostomy
* able to give informed consent as documented by signature

Exclusion Criteria:

* dementia or other psychiatric disorder that would prevent the patients from answering the questionnaires and experiencing sustainable training effects
* impossibility of stoma reversal due to persistent anastomotic leak and/or local recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of the LARS score after 13 months | 13 months after closure of ileostomy
  The primary outcome is the change of the LARS score after participation for 13 months in an intensified follow-up program compared to standard treatment which means patients are only treated if they present themselves in our consultation hours due to complaints. The LARS score is recorded using the LARS score questionnaire, developed 2012 by Emmertson et al.. The LARS score consists of five questions on the topics incontinence for flatus, incontinence for liquid stools, frequency of bowel movements, clustering of stools and urgency. Each answer results in a number of points, those points are summarized in the end to give a total score. This score is categorized into a range of no LARS (score 21 and lower), minor LARS (score 21 - 29) and major LARS (score 30 - 42).

SECONDARY OUTCOMES:
Patients' quality of life (QoL) | 1, 4, 7 and 13 months after closure of ileostomy
  Patients' quality of life will be recorded using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Colorectal Cancer (EORTC-QLQ-CR29) which will be filled out by the patients before closure of ileostomy as well as 1, 4, 7 and 13 months after closure of ileostomy.
  Maximum score is 140 points, minimum score 35 points. Higher scores mean worse outcomes.
Urinary symptoms in women and men | 1, 4, 7 and 13 months after closure of ileostomy
  Urinary symptoms in women and men will be recorded using the American Urological Association Symptom Index (AUA-SI) which is a validated questionnaire for urinary symptoms in women and men.
  Maximum score is 35 points, minimum score 0 points. Higher scores mean worse outcomes.
Sexual function in women | 1, 4, 7 and 13 months after closure of ileostomy
  Sexual function in women will be recorded using the International Consultation on Incontinence Questionnaire Female Sexual Matters Associated with Lower Urinary Tract Symptoms Module (ICIQ-FLUTSsex) which is a validated questionnaire for sexual complaints in women.
  Maximum score is 14 points, minimum score 0 points. Higher scores mean worse outcomes.
Sexual function in men | 1, 4, 7 and 13 months after closure of ileostomy
  Sexual function in men will be recorded using the International Index of Erectile Dysfunction (IIEF-5) which is a validated questionnaire for sexual complaints in men.
  Maximum score is 25 points, minimum score 5 points. Higher scores mean better outcomes.
Readmission to hospital | 13 months
Costs | 13 months
Compliance to treatment intervention | 13 months
  Recording of drop-outs, patients refusing to participate in interventions, tolerance of the medication and recording of side effects.
Natural history of incidence of LARS symptoms in control group | 13 months
  Incidence of LARS symptoms will be measured by the LARS score. The LARS score consists of five questions on the topics incontinence for flatus, incontinence for liquid stools, frequency of bowel movements, clustering of stools and urgency. Each answer results in a number of points, those points are summarized in the end to give a total score. This score is categorized into a range of no LARS (score 21 and lower), minor LARS (score 21 - 29) and major LARS (score 30 - 42).
Prevalence of LARS | 13 months
Rate of secondary ostomy formation | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Steinemann, Deputy chief physician, Study Chair — Clarunis - Universitäres Bauchzentrum Basel
Locations (5):
- Switzerland (5):
  - Clarunis Universitäres Bauchzentrum Basel, Basel
  - Lindenhofspital Bern, Bern
  - St. Anna Spital Bern, Bern
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Roberts RO, Jacobsen SJ, Jacobson DJ, Reilly WT, Talley NJ, Lieber MM. Natural history of prostatism: high American Urological Association Symptom scores among community-dwelling men and women with urinary incontinence. Urology. 1998 Feb;51(2):213-9. doi: 10.1016/s0090-4295(97)00505-0. PMID 9495700
- [Background] Rosen RC, Cappelleri JC, Smith MD, Lipsky J, Pena BM. Development and evaluation of an abridged, 5-item version of the International Index of Erectile Function (IIEF-5) as a diagnostic tool for erectile dysfunction. Int J Impot Res. 1999 Dec;11(6):319-26. doi: 10.1038/sj.ijir.3900472. PMID 10637462
- See also: Quality of life questionnaire (EORTC-QLQ-CR29 for colorectal cancer) — https://qol.eortc.org/questionnaires/
- See also: ICIQ-FLUTSsex (questionnaire for sexual complaints in women) — https://iciq.net/iciq-flutssex